CLINICAL TRIAL: NCT05528003
Title: Comparison of Homemade Versus Commercialized Single-access Port Devices for Single-incision Laparoscopic Appendectomy: A Retrospective Comparative Study
Brief Title: Homemade Versus Commercialized Single-access Port Devices in Single-incision Laparoscopic Appendectomy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202104032RINB
Record Dates: First submitted 2022-08-31; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Minimally Invasive Surgical Procedures
Keywords: Single-incision laparoscopic appendectomy; Single-access port device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Handmade single-access port device: The homemade single-access device was composed of a wound protector, sterile surgical glove, and three trocars inserted into and secured over three digits of the glove
- Commercialized single-access port devices: Commercialized single-access port devices including GelPOINT® (Applied Medical, Rancho Santa Margarita, CA, USA) and LAGIPORT® (LAGIS, Taichung, Taiwan)
  Interventions: Procedure: Commercialized single-access port devices

INTERVENTIONS:
Procedure: Commercialized single-access port devices — Two kinds of commercialized single-access port devices were used.
  Groups: Commercialized single-access port devices

SUMMARY:
Homemade and commercialized single-assess port devices are two kinds of port devices commonly used for single-incision laparoscopic appendectomy. This study aimed to compare these two port devices in terms of short-term surgical outcomes and medical costs.

DETAILED DESCRIPTION:
The advantages of homemade port devices include accessibility of the composites and lower equipment costs to the patients; however, the potential disadvantage is the easy leakage of CO2, ballooning of the surgical glove, and device instability, leading to difficult maneuverability. On the other hand, commercialized port devices have relatively easy maneuverability, flexibility for instrument changes, and port stability for long-duration surgery ; however, their higher equipment cost is a disadvantage.

ELIGIBILITY:
Inclusion Criteria:

* The patients were diagnosed as acute appendicitis and undergoing single-incision laparoscopic appendectomy

Exclusion Criteria:

* The patient was not diagnosed as acute appendicitis based on surgical finding or pathological findings
* The patients underwent surgery other than single-incision laparoscopic surgery

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute appendicitis patients
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Total surgical complications | Complications happened within 30 days
  Complications were defined by Clavien-Dindo classification and comprehensive complication index.
Superficial incisional surgical site infection (SSI) | Complications happened within 30 days
  SSI was defined according to the American Centers for Disease Control and Prevention (CDC) classification
Deep/organ SSI | Complications happened within 30 days
  SSI was defined according to the American Centers for Disease Control and Prevention (CDC) classification
Postoperative ileus | Complications happened within 30 days
  Postoperative ileus was defined as the presence of symptoms and signs of abdominal distention, nausea, or vomiting combined with abdominal radiography, such as plain radiography or CT, within 30 days after SILA.

SECONDARY OUTCOMES:
Surgical time | Time from skin incision to application of gauzes
  Total time needed for completing surgery
Time to resume soft diet | The time to resume a soft diet was measured as the duration between the time leaving the recovery room and the time to resume a soft diet recorded in the nursing note.
  Total time needed to resume bowel ability to resuming soft diet
Postoperative length of hospitalization | Postoperative LOH was defined as the duration between leaving the recovery room and discharge.
  Total time to stay in hospital
Total medical costs | From the time patient being brought to emergency room to the time patient being discharged
  Medical costs were defined as the medical fees paid by the National Health Insurance and did not include the self-paid equipment fees needed in SILA (e.g., commercialized single-access port devices, or wound protector).

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Tso LIAO, MD, Principal Investigator — NTUH, Hsin-Chu Hospital

IPD SHARING:
Plan to Share IPD: No